EduCan Trial: Study protocol for a randomized controlled trial on the effectiveness of Pain Neuroscience Education after breast cancer surgery on

pain-, physical-, emotional- and work-related functioning

Trial Registration: ClinicalTrials.gov Identifier: NCT03351075

Ethical Committee of the University Hospitals Leuven: s60702

Document date: august 2024

1

#### **INTRODUCTION**

Breast cancer is the most frequent malignancy among women worldwide. (1) Despite the high incidence, in Western countries an increase in survival and life expectancy has been observed due to the ongoing improvement of detection method accuracy, early diagnosis, and breast cancer treatment.(1) Consequently, more attention is warranted towards the debilitating problems accompanying this disease and its treatment, which can persist for months or even years after diagnosis. In addition to fatigue, pain is the most frequent and persistent symptom following cancer and cancer treatment. Between 27 and 79% of women report pain one month after surgery, which is often attributed to local pain mechanisms caused by a postsurgery and/or radiotherapy tissue insult at that time-point. (2-5) One would expect prevalence rate to diminish as healing occurs, yet this does not seem to be the case. In fact, 12-82% of women still report persistent pain one year or later.(4) This may indicate that besides local nociceptive and neuropathic pain mechanisms, a third pain mechanism characterized by altered nociceptive processing without clear evidence of persistent tissue damage causing the activation of peripheral nociceptors (i.e. nociceptive pain) or evidence for disease or lesion of the somatosensory system causing the pain (i.e. neuropathic pain). (17-19) Moreover, pain interferes with pain-, physical-, emotional- and work-related disability and therefore severely prejudices a person's quality of life (QOL) and participation in society.(6-8) Hence, adequate pain management in the early stage of breast cancer treatment is necessary to prevent and improve pain and pain-related disability, both at short- and longterm.

Despite the effectiveness of currently applied physical therapy modalities after breast cancer surgery (such as manual techniques, specific exercises and general exercises), up to 72% of women still experience pain and the resulting disabilities after finishing breast cancer treatment.(9) Over the past decades, awareness on the important role of educational interventions in the management of cancer pain has increased.(10-12) These general educational interventions have been shown to be effective for improving pain severity, self-efficacy and knowledge and attitude to pain and analgesia in cancer patients. However, effect sizes are only moderate and of limited clinical relevance.(10) This can be explained by the fact that these educational interventions mainly focus on tissue and tissue injury as the source of

pain and are often restricted to biomedical pain management instructions and general advice on physical activity and analgesics.(10-12) They focus on explaining treatment side-effects and improving patients' coping strategies. Recently, increased knowledge on pain mechanisms has led to a more modern educational approach, also known as Pain Neuroscience Education (PNE).(13-16) This explains the neurophysiology of chronic pain and the ability of the nervous system to modulate pain experience, as well as the potential influences of sleep, thoughts, feelings and culture, among others, on pain. Thereby, it targets a reconceptualization from a biomedical or structural model to an actual biopsychosocial model of pain. Through the knowledge that pain is often an unreliable indicator of the presence or extent of tissue damage and if patients may become open to exploring broader contributions to pain, pain-related behavior might change by shifting from passive therapyreceiving to active self-management. Increased knowledge of the broad contributions to pain (4), as well as awareness of different pain mechanisms following breast cancer treatment (17-19) provides justification for the integration of PNE in this population. Applying PNE could enhance the effectiveness of the currently applied physical therapy modalities for prevention and treatment of pain and related disabilities after breast cancer treatment, compared to a traditional biomedical educational intervention. Indeed, encouraging people to address emotional, cognitive and broader health-related factors in the early stage of cancer treatment may enhance recovery during and after the treatment. To our knowledge, only one controlled trial investigated the effectiveness of PNE in the early stage of breast cancer treatment.(20) Although the results were very promising for shoulder function, only short-term effects were examined, no randomization was performed and no pain-related or other health-related outcomes were evaluated.

### **Objectives**

The main scientific objective is to examine the effectiveness of PNE, in addition to a standard best evidence physical therapy program, on pain-, physical-, emotional-, and work-related functioning in the early stage of breast cancer treatment, compared to a traditional biomedical educational intervention, up to 1.5 years after surgery (EduCan Trial). This will be performed through a double-blinded randomized controlled trial.

# **METHODS AND ANALYSIS**

Described according to the SPIRIT guidelines (http://www.spirit-statement.org/protocol-version/).

# Trial design and study setting

A parallel, two-arm randomized controlled trial with blinding of assessors and physical therapists providing the standard physical therapy program in both arms and masking of the participants. The trial started in November 2017 at the department of Physical Medicine and Rehabilitation of the University Hospitals in Leuven (Belgium). A schedule of the EduCan Trial is provided in Table 1.

Table 1. Schedule of enrolment, interventions, and assessments of the EduCan Trial

| | STUDY PERIOD | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Enrolment | | Allocati<br>on | Post-allocation | | | | |
| TIMEPOINT | <b>-t</b> <sub>2</sub><br>preop<br>consult | - <b>t</b> <sub>1</sub><br>postop<br>consult | 0 | <b>t</b> <sub>1</sub><br>4 Mo | <b>t</b> <sub>2</sub><br>6 Mo | <b>t</b> ₃<br>8 Mo | t <sub>4</sub><br>12 Mo | <b>t</b> 5<br>18 Mo |
| ENROLMENT | | | | | | | | |
| Eligibility screen | X | | | | | | | |
| Informed consent | Х | | | | | | | |
| Randomization | | | х | | | | | |
| Allocation | | | Х | | | | | |
| | | INT | ERVENTI | ONS | | | | |
| | | | | Intensive<br>phase | Ма | | | |
| Standard PT program (All) | | n=184 | | 1-2<br>sessions<br>/week | 1<br>session | 1<br>session | 1<br>session | |
| Pain Neuroscience<br>Education (IG) | | n=92 | | 3<br>sessions | 1<br>session | 1<br>session | 1<br>session | |
| Biomedical Education (CG) | | n=92 | | 3<br>sessions | 1<br>session | 1<br>session | 1<br>session | |
| ASSESSMENTS | | | | | | | | |
| Pain-related functioning (primary outcome)* | Х | Х | | Х | Х | Х | Х | Х |
| Pain-related outcomes* | Х | Х | | Х | Х | Х | Х | Х |
| Emotional functioning | Х | Х | | Х | Х | Х | Х | Х |
| Physical functioning* | | Х | | Х | | | Х | Х |
| Work-related functioning* | | | | х | Х | Х | Х | Х |

<sup>\*</sup>see Table 2 for details on the content of the different assessments at each point in time Mo = Months; IG=Intervention Group; CG=Control Group

### Patient and public involvement in trial design

One female breast cancer patient and a representative of the National Health Service were consulted during the initial grant preparation and trial set up. The patient representative provided valuable insight into the worries and concerns experienced during cancer treatment. The representative of the National Health service contributed to the design of the study and advised on assessment of work-related functioning outcomes.

### **Eligibility criteria**

Women are eligible to participate in the EduCan Trial if they are scheduled for surgery for breast cancer at the Multidisciplinary Breast Center of the University Hospitals of Leuven. Patients with increased risk of developing pain after breast cancer surgery are included.(21-23) Therefore, inclusion criteria are: 1) diagnosed with histologically confirmed invasive or non-invasive primary breast cancer, 2) scheduled for surgical excision including either axillary lymph node dissection and mastectomy (whether or not in combination with reconstructive surgery) or breast-conserving; or either sentinel node biopsy and mastectomy (whether or not in combination with reconstructive surgery); 3) aged 18 years or older; 4) can comply with the study protocol. Patients with active metastasis are excluded because of the higher risk of mortality.

### Participant screening, recruitment and consent.

Participants are identified from scheduled operation lists and screened for eligibility criteria. The initial screening process is undertaken by a member of the research team. Potentially eligible participants are approached and recruited during the *preoperative consult* at the Multidisciplinary Breast Center of the University Hospitals of Leuven. All eligible patients receive an information sheet and the explanation of the study during the preoperative consult. Next, they are asked to have a preoperative baseline measurement for which a separate informed consent exists. Because of ethical and deontological reason patients will not be forced to decide on participation in the complete EduCan Trial at this moment, but initially only for the baseline measurements.

During their *postoperative hospital stay*, a member of the research team will meet the eligible participants again, answer further questions and include them in the further trial if wanted.

Then, a second informed consent is signed for participating in the complete EduCan Trial. The preoperative baseline measurement of non-participating patients will be stored in the medical file of the patient and can be consulted on clinical follow-up appointments to evaluate the recovery of the patient but is not used for research purpose. The participants' flow is summarized in Figure 1.

Figure 1: Flow diagram of the EduCan Trial



<sup>\*</sup>A separate informed consent is available for the preoperative assessment Mo=Months

#### Allocation and randomization

Therapists and assessors are blinded to the allocation of the treatment groups. The therapists providing the standard physical therapy program will be unaware of the type of education received by the patient (PNE in the intervention group and biomedically-focused education in the control group). Assessors are blinded to the maximal extent possible. With regard to this, patients are asked not to communicate with the assessors about the intervention

received. Patients are masked for the allocation to the intervention/control group; they do not know which one is the experimental intervention and which one is the control intervention, however they will of course be aware of the intervention received.

At the end of the trial, the success of assessor blinding will be examined by asking whether the assessor thought the participant had received the experimental or control intervention, including the percentage of certainty (i.e. 50% certainty means a pure guess). The same will be done for patient masking. The research members performing statistical analysis will be blinded as well.

The randomization is computer-generated and is performed by using permuted blocks (size=4). An independent co-worker at the department carries out the randomization to ensure blinding of the research team. The sequence of randomization is determined by the patient's identification number, which she receives after signing informed consent. Participants are randomized in a 1:1 ratio between intervention and control arms.

#### **Interventions**

Standard physical therapy program

All participants in the EduCan Trial attend a standard physical therapy program. The standard physical therapy program is based on currently available evidence and clinical experience of the research team and will include three physical therapy modalities. First, **manual techniques** including (a) passive mobilizations to restore shoulder range of motion, (b) stretching of the pectoral muscles to improve muscle flexibility and (c) scar tissue massage to improve flexibility of the scar(s) will be implemented. (9, 24, 25) Second, **specific exercises** to improve shoulder range of motion and upper limb strength have been proven to be effective for treatment of upper limb problems after breast cancer and will start immediately after surgery as well. (9, 26) Specific exercises are instructed during the individual session and continued at home. Third, patients are advised on **general exercises**. General exercises should be implemented to increase patient's physical activity level. In general, these recommendations consist of physical activity at a minimum level of moderate intensity over an extended period and can include e.g. running, walking, cycling, swimming, etc. (27, 28)

During month 1-4 an **intensive physical therapy program** is implemented because of the postoperative side-effects. Patients will attend 1-2 individual sessions of 30 minutes per week

during the intensive phase, starting one week post-surgery. All patients start with a frequency of two sessions per week, decreasing to once each two weeks. The decrease in frequency of the sessions is pragmatically chosen based on the individual progression and need of the patient.

Up to one year after surgery a **maintenance physical therapy program** is implemented to follow-up on the exercises performed at home and to treat possible additional/ new side-effects of other adjuvant treatment modalities such as radiotherapy, chemotherapy and hormone therapy. An individual maintenance session of 30 minutes is scheduled 6, 8 and 12 months post-surgery.

Additionally, **information about prevention of lymphedema** is given by a specialized physical therapist: about normal use of the upper limb, avoiding pinching off the arm, skin care and control of body weight.(29) One group information sessions of 60 minutes on this topic is organised each month which should be attended once by every participant (both patients from the intervention and control group together) and this as soon as possible after surgery. Patients also receive a brochure with this information. If patients develop lymphedema they are additionally referred to the Lymfovenous Center of the University Hospitals of Leuven for further treatment of the lymphedema.

#### Educational intervention

The educational sessions are individual and last for 30 minutes. The first PNE session is given within the first postoperative week before the start of the standard physical therapy program to prepare the patient for the physical therapy sessions. Information is presented verbally (explanation by the therapist) and in multi-media forms (power point presentation with summaries, pictures, metaphors and diagrams on computer). After the first session, patients also receive an information leaflet on paper and are asked to read it carefully at home. They also receive a web-link to an online presentation that summarizes the provided information. Additional written information that can be read afterwards is a valuable and essential part of the educational intervention. In the following 4 weeks after surgery, 2 additional PNE sessions are provided to ensure that the patient understands the pain physiology and principles of activity management and can relate this to the physical therapy program and his/her pain complaint. However, education is a continuous process initiated at the start and continuing

into and followed-up during the longer-term rehabilitation program. Therefore, three additional booster sessions are organized at 6, 8 and 12 months post-surgery. During the booster sessions, the information given postoperatively will be rehearsed and application of the information into future stages of the recovery process will be discussed. Special attention is given to return to preoperative activities and return to work (if applicable). Regarding this, a second information leaflet on paper will be given to the patient. Patients in the control arm and intervention arm will have the same schedule of educational sessions, only the content of the education differs from the intervention arm.

### Intervention arm: Pain Neuroscience Education (PNE)

Based on the available literature a modern PNE program has been established to *explain pain* specifically for this population.(10, 12, 20) The content and pictures of the educational sessions are based on the book 'Explain Pain' (Butler & Moseley, 2003), 'Pijneducatie een praktische handleiding voor (para)medici' (Van Wilgen & Nijs, 2011) and the 'The Pain Toolkit' (Peter Moore, 2002), as used in earlier studies.(30, 31) Topics addressed during the PNE sessions will include: the characteristics of acute versus chronic pain; specific side effects of the different breast cancer treatment modalities in relation to pain; how pain is a product of the brain; how pain becomes chronic (plasticity of the nervous system, modulation, modification, central sensitization); potential sustaining factors of pain such as emotions, stress, pain cognitions, and pain behavior.

Additionally, this PNE intervention includes advice for *activity management*, while experiencing pain and other symptoms. In addition to the general recommendations for general exercise and advice to stay active in the standard physical therapy program, the PNE guides patients in performing general exercises and activities according to the graded activity principle. Graded activity is applied according to the guidelines reported by the International Association for the Study of Pain (IASP).(32) This includes general exercise activities according to pacing strategies for 'persisters' (i.e. restructuring the activity pattern to avoid peaks of over activity and exacerbations of their pain) and graded activity for 'avoiders' (i.e. time-contingent increase of physical activity). PNE is crucial here to help patients interpret pain during exercise in the correct context. Finally, advice on *returning to work* in the context of present pain complaints and how to apply the principles described above for activity management can be applied in the working situation will be provided.

Control arm: Traditional biomedical education

Traditional biomedical educational interventions consist of explaining patient's pain experience in relation to the therapeutic procedures from a tissue and biomechanical perspective.(33, 34) Information on the different side effects of surgery, radiotherapy, chemotherapy, hormone therapy and target therapy is given. The role of different structures and injured versus healthy tissue in acute and persistent pain is discussed. Pain is explained from a biomechanical point of view, e.g. deviance from normal expected movement patterns and postures. Additionally, during the educational sessions and rehabilitation program, patients receive advice on activity management. This advice is to stay active as minimally possible during treatment and increase their physical activity level according to current recommendations for general exercises after treatment. Based on the American Cancer Society Guidelines on Physical Activity at least 150 minutes of moderate intensity (heart rate 50 to 70% of the maximum heart rate or a score of 12-14 on Borg Rating of Perceived Exertion (RPE)) or 75 minutes of vigorous intensity activity (70 to 85% of the maximum heart rate or RPE of > 15) each week (or a combination of these), preferably spread throughout the week is recommended. Finally, advice on returning to work in the context of the different (persistent) side-effects of the treatments will be provided.

#### Outcomes

The outcome measures were chosen in accordance with the guideline for **core outcome domains** to be used in clinical trials on multimodal treatment approaches for pain as advocated by an international steering committee (**VAPAIN recommendations**)(35) and the **IMMPACT recommendations** for the outcome measures in pain clinical trials.(36)

The primary outcome is pain-related functioning at 12 months measured using the Pain Disability Index (PDI). Secondary outcomes are other pain symptoms and characteristics, physical functioning, emotional functioning and work-related functioning. Assessments are performed within one week preoperatively, within one week postoperatively and then at 4 months, 6, 8, 12 and 18 months after surgery. However, because of feasibility limitations not all outcome parameters are assessed at each assessment time point. Table 1 and 2 present the study outcome measures by assessment time point. In table 3 the outcome measures are described in more detail.

Table 2. Study outcome measures by assessment time point

| Domain | Scale/measure | T <sub>-2</sub><br>1W<br>preop | T <sub>-1</sub><br>1W<br>postop | T <sub>1</sub><br>4 Mo | T <sub>2</sub><br>6 Mo | T <sub>3</sub><br>8 Mo | T <sub>4</sub><br>12<br>Mo | T₅<br>18<br>Mo |
|---|---|---|---|---|---|---|---|---|
| Pain-related<br>functioning<br>(primary<br>outcome) | Pain Disability Index | х | х | х | х | х | х | х |
| Pain | Pain intensity (VAS) | Х | Х | Х | Х | Х | х | Х |
| symptoms | Brief Pain Inventory (BPI) | Х | Х | Х | Х | Х | Х | Х |
| and characteristics | Neuropathic Pain Questionnaire (DN4) | X | Х | Х | Х | Х | Х | x |
| | Central Sensitisation Questionnaire (CSI) | х | х | Х | Х | Х | х | х |
| | Pain sensitivity testing | Х | Х | Х | Х | Х | х | Х |
| Physical functioning | General physical activity level (accelerometry) | | Х | Х | | | х | х |
| | Upper limb performance (accelerometry) | | х | Х | | | х | Х |
| | Upper limb function (DASH) | Х | Х | Х | Х | Х | Х | Х |
| Emotional functioning | Pain Catastrophizing Scale (PCS) | X | Х | Х | Х | Х | Х | x |
| | Depression, Anxiety and Stress<br>Scale (DASS-21) | х | Х | Х | Х | Х | Х | х |
| | Health-related quality of life (McGill Quality of life questionnaire) | Х | х | х | х | х | Х | Х |
| Social | Return to work rate | | | х | Х | Х | Х | Х |
| functioning | QuickScan | | | Х | Х | Х | Х | Х |
| | Return-to-work self-efficacy (RTWSE-19) | | | Х | Х | Х | Х | Х |

Table 3. Outcome measures of the EduCan Trial

| Outcome | Assessment method |
|---|---|
| PAIN-RELATED FUNCTIONING (prima | ry outcome) |
| Pain-related functioning | Pain Disability Index (PDI). The PDI is a short, self-reported questionnaire for measuring the degree of interference of pain with normal role functioning (family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activity).(37, 38) |
| PAIN SYMPTOMS AND CHARACTERIS | TICS |
| Pain intensity | Visual Analogue Scale (VAS). Present pain intensity and mean pain intensity during the past week for pain at the upper limb region (i.e. shoulder-neck region, arm, axilla, trunk side and breast region) |
| Brief Pain Inventory | Medication use, pain quality, pain location, pain severity and response to treatment.(39) |
| Presence of neuropathic pain | Douleur Neuropathique en 4 questions (DN4). The DN4 a questionnaire generating reliable and valid data for identifying pain of predominantly neuropathic origin.(40) |
| Presence of hypersensitivity of the central nervous system | Central Sensitisation Inventory (SCI). The CSI is a questionnaire generating reliable and valid data to assess symptoms related to central sensitization mechanisms.(41) |
| Pain sensitivity testing - Quantitative Sensory testing: Mechanical detection and pain thresholds* | Twelve monofilaments (MARSTOCK nerve test - Optihair2, Schriesheim, Germany) with a force from 0.25 to 512 mN are used. The mechanical detection threshold is defined as the lowest mechanical force that the participant can detect. The mechanical pain threshold is defined as the lowest mechanical force that the participant perceives as painful or unpleasant. Monofilaments are applied with a rate of 2 seconds 'on' and 2 seconds 'off' at the inner side of the upper arm and lateral trunk side. |
| - Quantitative Sensory testing:<br>Temperature detection and pain<br>thresholds* | The computerized thermotest device TSA-II-NeuroSensory Analyser is used. The method of limits is used. The detection and pain thresholds are measured as the first identified stimulus under increasing stimulus intensities. The participant has to push the button once the stimulus is detected or perceived as painful or unpleasant. This is repeated three times for each threshold. The mean of three stimuli for each threshold is calculated and used for analysis.(42). |
| - Quantitative Sensory testing:<br>Pressure Pain Thresholds* | Measured by a digital Wagner FPX™ algometer. Points of measurement are defined by palpation for most tender muscle points (one per muscle) at the major pectoral muscle region, the lateral trunk side and upper trapezius muscle region. The participant is asked to say 'stop' when the sensation of pressure first changes to pain. The mean value of the 2 measurements is calculated and used for analysis.(43) |
| <ul> <li>Presence of widespread<br/>pain/secondary hyperalgesia</li> </ul> | Quantitative Sensory Testing is performed both at the local painful area as at remote body parts (i.e. quadriceps muscle at the nonaffected side) and pain distribution is displayed on a body diagram |
| - Presence and degree of impaired nociceptive inhibitory | Assessment of conditioned pain modulation will be done using the Medoc two thermode Q-Sense CPM system. This system involves a 'test' stimulus and a 'conditioning' stimulus applied on the ulnar |

| mechanisms (i.e. conditioned pain modulation) | side of the forearms. The test stimulus (at the affected side) is used to assess pain sensitivity to a warmth stimulus pre- and post the noxious conditioning stimulus and the difference is calculated between pre- and post-measures. When the second pressure pain threshold (i.e. test stimulus) is similar or lower than the first, dysfunctional inhibitory pain mechanisms are present. (44, 45) |
|---|---|
| - Presence and degree of<br>enhanced facilitation mechanisms<br>(i.e. wind-up) | Wind-up of pain or temporal summation will be assessed by applying repetitive nociceptive stimulation with a 26g Nylon monofilament at the major pectoral muscle at the affected side. The perceived intensity of the stimulus (the first, the last and aftersensations) are reported by using a Numeric Rating Scale. The temporal summation value is calculated as the difference between the first and the last stimuli or the slope of the increase in pain intensity. A response for enhanced temporal summation is deemed positive if participants perceive the initial stimulus as non-noxious, but it becomes noxious, increasing by at least two-points on a Numeric Rating Scale, or if baseline pain intensity increases by at least two points. (44-46) |
| - Presence and degree of | The Central Sensitization Inventory, a questionnaire generating |
| hypersensitivity to non- | reliable and valid data to assess symptoms related to central |
| mechanical stimuli | sensitization mechanisms (47-49) |
| PHYSICAL FUNCTIONING | |
| General physical activity and upper | Three ActiLife accelerometers, one on the pelvis (7 consecutive |
| limb performance | days) and one on each wrist (3 consecutive days), will be worn during waking hours. Outcome parameters are general activity level, unimanual/bimanual time and intensity of both unimanual/bimanual use. The ActiLife v6.9.5 Firmware v2.2.1 will be used to save raw data. Data will be further processed with Matlab®, using custom-written routines.(50, 51) |
| Upper limb function | DASH questionnaire. The DASH is a self-reported questionnaire on upper limb function.(3) |
| EMOTIONAL FUNCTIONING | |
| Pain catastrophizing | Pain Catastrophizing scale (PCS). The PCS is a self-reported |
| | questionnaire measuring catastrophic thinking related to pain. (53) |
| Depression, anxiety and stress | Depression Anxiety Stress scales 21 (DASS-21). The DASS-21 is a self-reported questionnaire that measures the three related states of depression, anxiety and stress. (54) |
| Health-related quality of life | McGill Quality of Life questionnaire (55) |
| SOCIAL FUNCTIONING | |
| Return to work rate | Self-reported questionnaire on return to work, employment status, work adjustments |
| QuickScan | Questionnaire on health status and return-to-work obstacles in order to assess potential predictive factors for long-term absenteeism. |
| Patients perceived ability to work | Return-to-work self-efficacy questionnaire (RTWSE-19). The RTWS 19 is a self-reported questionnaire on the patients' perceived abilit to work.(56) |
| * Testing is performed hilaterally, exce | pt preoperatively because of feasibility reasons |

<sup>\*</sup> Testing is performed bilaterally, except preoperatively because of feasibility reasons

# Sample size

A power calculation was performed by the Leuven Biostatistics and statistical bioinformatics Centre of KU Leuven for the primary outcome parameter 'Pain Disability Index (PDI) after 1 year". Sample size calculation was based on data available in literature for the PDI.(37, 38) and calculated to detect with 80% power a difference of 20% in Pain Disability Index after 1 year. Assuming a coefficient of variation (CV) equal to 0.5, 87 participants per group are needed based on a two-sample pooled t-test of a mean ratio with lognormal data and setting alpha equal to 0.05. The assumed CV is a conservative estimate, derived from the observed CV of 0.30 in a sample of normative data for women with chronic pain. To anticipate a dropout rate of approximately 5%, 184 participants in total will be recruited. The drop-out rate is based on previous similar trials at our institution.(29, 57, 58) To handle the potential missing measurements after 1 year, the comparison of the PDI will be based on a multivariate normal model for longitudinal measurements fitted on all repeated measures over time (pre-op, postop, 4, 6, 8, 12 and 18 months). A log-transformation will be applied if necessary to handle the right-skewed distribution of the PDI.

### **Data analysis**

Statistical analysis will be intention-to-treat and will comply with the Consolidated Standards of Reporting Trials (CONSORT) guidelines. Analysis will be conducted in a blinded way. The continuous data will be summarized using mean, SD, median and range values. The primary outcome will be analyzed using multilevel linear regression models for repeated (longitudinal) measures, using an unstructured covariance matrix. The mean change from baseline (i.e. preoperative assessment) to 4, 6, 8, 12 and 18 months (with correction for the postoperative assessment), will be estimated using contrast statements for each of the treatment arms. The difference in mean changes and their 95% CIs between interventions will be plotted graphically so that change can be assessed over the course of the study. Continuous secondary outcomes will be assessed in a similar way to the primary outcome. Categorical data will be analyzed using logistic models. For non-repeated continuous and binary measurements, ordinary linear regression and logistic models will be used, respectively.

#### Data security and management

Participant data are stored on a secure database in accordance with the General Data Protection Regulations (2018). Data is de-identified and a unique trial identification number

used on all participant communication. Clinical and patient forms are being checked for completeness and congruity before data entry onto the database. Data will undergo additional checks to ensure consistency between data submitted and original paper forms. Trial documentation and data will be archived for at least 10 years after completion of the trial.

# **Trial monitoring**

The steering committee of the research team will oversee all aspects of design, delivery, quality assurance and data analysis. The steering committee will monitor the trial at least once per year.

### **ETHICS AND DISSEMINATION**

#### **Ethical considerations**

The EduCan Trial applies the principles established in the Declaration of Helsinki. Participants provide written informed consent before data collection. Only de-identified coded and interpreted data will be shared between the members of the research team. Ethics approval was granted by the local Ethical Committee of the University Hospitals Leuven (s60702).

#### **Dissemination of results**

The research team are committed to full disclosure of the results of the trial. Findings will be reported in accordance with CONSORT guidelines and we aim to publish in high impact journals. Given the multitude of outcome parameters, results will be divided over several papers. Our patient representatives and representative of the National Health Service will assist with dissemination of study results. The funder will take no role in the analysis or interpretation of trial results.

# Acknowledgements

The authors would like to thank all the trial participants. The authors would also like to thank all the physical therapy staff, surgical oncology teams, breast cancer nurses and research departments collaborating on this study.

#### **REFERENCES**

- 1. Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, et al. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. International journal of cancer Journal international du cancer. 2015;136(5):E359-86.
- 2. Rietman JS, Dijkstra PU, Geertzen JH, Baas P, De Vries J, Dolsma W, et al. Short-term morbidity of the upper limb after sentinel lymph node biopsy or axillary lymph node dissection for Stage I or II breast carcinoma. Cancer. 2003;98(4):690-6.
- 3. Hidding JT, Beurskens CH, van der Wees PJ, van Laarhoven HW, Nijhuis-van der Sanden MW. Treatment related impairments in arm and shoulder in patients with breast cancer: a systematic review. PloS one. 2014;9(5):e96748.
- 4. Wang L, Guyatt GH, Kennedy SA, Romerosa B, Kwon HY, Kaushal A, et al. Predictors of persistent pain after breast cancer surgery: a systematic review and meta-analysis of observational studies. Cmaj. 2016;188(14):E352-e61.
- 5. Leysen L, Beckwee D, Nijs J, Pas R, Bilterys T, Vermeir S, et al. Risk factors of pain in breast cancer survivors: a systematic review and meta-analysis. Supportive care in cancer: official journal of the Multinational Association of Supportive Care in Cancer. 2017.
- 6. Kudel I, Edwards RR, Kozachik S, Block BM, Agarwal S, Heinberg LJ, et al. Predictors and consequences of multiple persistent postmastectomy pains. Journal of pain and symptom management. 2007;34(6):619-27.
- 7. Sun Y, Shigaki CL, Armer JM. Return to work among breast cancer survivors: A literature review. Supportive care in cancer: official journal of the Multinational Association of Supportive Care in Cancer. 2017;25(3):709-18.
- 8. Shin WK, Song S, Jung SY, Lee E, Kim Z, Moon HG, et al. The association between physical activity and health-related quality of life among breast cancer survivors. Health and quality of life outcomes. 2017;15(1):132.
- 9. De Groef A, Van Kampen M, Dieltjens E, Christiaens MR, Neven P, Geraerts I, et al. Effectiveness of postoperative physical therapy for upper-limb impairments after breast cancer treatment: a systematic review. Archives of physical medicine and rehabilitation. 2015;96(6):1140-53.
- 10. Bennett MI, Bagnall AM, Jose Closs S. How effective are patient-based educational interventions in the management of cancer pain? Systematic review and meta-analysis. Pain. 2009;143(3):192-9.
- 11. Armes J, Chalder T, Addington-Hall J, Richardson A, Hotopf M. A randomized controlled trial to evaluate the effectiveness of a brief, behaviorally oriented intervention for cancer-related fatigue. Cancer. 2007;110(6):1385-95.
- 12. Ling CC, Lui LY, So WK. Do educational interventions improve cancer patients' quality of life and reduce pain intensity? Quantitative systematic review. Journal of advanced nursing. 2012;68(3):511-20.
- 13. Moseley GL, Butler DS. Fifteen Years of Explaining Pain: The Past, Present, and Future. The journal of pain: official journal of the American Pain Society. 2015;16(9):807-13.
- 14. Nijs J, Meeus M, Van Oosterwijck J, Roussel N, De Kooning M, Ickmans K, et al. Treatment of central sensitization in patients with 'unexplained' chronic pain: what options do we have? Expert opinion on pharmacotherapy. 2011;12(7):1087-98.

- 15. Nijs J, Paul van Wilgen C, Van Oosterwijck J, van Ittersum M, Meeus M. How to explain central sensitization to patients with 'unexplained' chronic musculoskeletal pain: practice guidelines. Manual therapy. 2011;16(5):413-8.
- 16. Nijs J, Torres-Cueco R, van Wilgen CP, Girbes EL, Struyf F, Roussel N, et al. Applying modern pain neuroscience in clinical practice: criteria for the classification of central sensitization pain. Pain physician. 2014;17(5):447-57.
- 17. Nijs J, Leysen L, Adriaenssens N, Aguilar Ferrandiz ME, Devoogdt N, Tassenoy A, et al. Pain following cancer treatment: Guidelines for the clinical classification of predominant neuropathic, nociceptive and central sensitization pain. Acta oncologica. 2016;55(6):659-63.
- 18. Nijs J, Leysen L, Pas R, Adriaenssens N, Meeus M, Hoelen W, et al. Treatment of pain following cancer: applying neuro-immunology in rehabilitation practice. Disability and rehabilitation. 2016:1-8.
- 19. De Groef A MM, Van der Gucht E, Dams L, Van Kampen M, Geraerts I, Devoogdt N. Unraveling self-reported signs of central sensitization in breast cancer survivors with upper limb pain: prevalence rate and contributing factors. Pain physician. 2017; *Accepted*.
- 20. Sato F, Ishida T, Ohuchi N. The perioperative educational program for improving upper arm dysfunction in patients with breast cancer: a controlled trial. The Tohoku journal of experimental medicine. 2014;232(2):115-22.
- 21. Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. The journal of pain: official journal of the American Pain Society. 2011;12(7):725-46.
- 22. De Groef A, Van Kampen M, Tieto E, Schonweger P, Christiaens MR, Neven P, et al. Arm lymphoedema and upper limb impairments in sentinel node-negative breast cancer patients: A one year follow-up study. Breast. 2016;29:102-8.
- 23. Katz J, Poleshuck EL, Andrus CH, Hogan LA, Jung BF, Kulick DI, et al. Risk factors for acute pain and its persistence following breast cancer surgery. Pain. 2005;119(1-3):16-25.
- 24. De Groef A, Van Kampen, M., Vervloesem, N., Dieltjens, E., Christiaens, MR., Neven, P., Geraerts, I, Devoogdt, N. Effect of myofascial techniques for treatment of persistent upper limb pain after breast cancer treatment: randomized controlled trial. *Submitted* . 2016.
- 25. De Groef AVK, M. Vervloesem, N. De Geyter, S. Christiaens, MR. Neven, P. Geraerts, I. Devoogdt, N. Myofascial techniques have no additional beneficial effects to a standard physical therapy program for upper limb pain after breast cancer surgery: a randomized controlled trial

. 2016.

- 26. McNeely ML, Campbell K, Ospina M, Rowe BH, Dabbs K, Klassen TP, et al. Exercise interventions for upper-limb dysfunction due to breast cancer treatment. Cochrane database of systematic reviews (Online). 2010(6):CD005211.
- 27. Zeng Y, Huang M, Cheng AS, Zhou Y, So WK. Meta-analysis of the effects of exercise intervention on quality of life in breast cancer survivors. Breast cancer. 2014.
- 28. Mishra SI, Scherer RW, Geigle PM, Berlanstein DR, Topaloglu O, Gotay CC, et al. Exercise interventions on health-related quality of life for cancer survivors. Cochrane database of systematic reviews (Online). 2012;8:Cd007566.
- 29. Devoogdt N, Christiaens MR, Geraerts I, Truijen S, Smeets A, Leunen K, et al. Effect of manual lymph drainage in addition to guidelines and exercise therapy on arm lymphoedema related to breast cancer: randomised controlled trial. BMJ (Clinical research ed). 2011;343:d5326.

- 30. Moseley L. Combined physiotherapy and education is efficacious for chronic low back pain. The Australian journal of physiotherapy. 2002;48(4):297-302.
- 31. Van Oosterwijck J, Meeus M, Paul L, De Schryver M, Pascal A, Lambrecht L, et al. Pain Physiology Education Improves Health Status and Endogenous Pain Inhibition in Fibromyalgia: A Double-Blind Randomized Controlled Trial. The Clinical journal of pain. 2013.
- 32. Mira Meeus JN, Paul van Wilgen, Suzie Noten, Dorien Goubert, Ivan Huijen. Moving on to Movement in Patients with Chronic Joint Pain. Pain Clinical Updates. 2016.
- 33. Louw A, Puentedura EJ, Zimney K, Schmidt S. Know Pain, Know Gain? A Perspective on Pain Neuroscience Education in Physical Therapy. Journal of Orthopaedic & Sports Physical Therapy. 2016;46(3):131-4.
- 34. Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiotherapy theory and practice. 2016;32(5):332-55.
- 35. Kaiser U, Kopkow C, Deckert S, Neustadt K, Jacobi L, Cameron P, et al. Developing a core outcome-domain set to assessing effectiveness of interdisciplinary multimodal pain therapy: the VAPAIN consensus statement on core outcome-domains. Pain. 2017.
- 36. Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, et al. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005;113(1-2):9-19.
- 37. Soer R, Reneman MF, Vroomen PC, Stegeman P, Coppes MH. Responsiveness and minimal clinically important change of the Pain Disability Index in patients with chronic back pain. Spine. 2012;37(8):711-5.
- 38. Chibnall JT, Tait RC. The Pain Disability Index: factor structure and normative data. Archives of physical medicine and rehabilitation. 1994;75(10):1082-6.
- 39. Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Annals of the Academy of Medicine, Singapore. 1994;23(2):129-38.
- 40. Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, et al. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005;114(1-2):29-36.
- 41. Kregel J, Vuijk PJ, Descheemaeker F, Keizer D, van der Noord R, Nijs J, et al. The Dutch Central Sensitization Inventory (CSI): Factor Analysis, Discriminative Power, and Test-Retest Reliability. The Clinical journal of pain. 2016;32(7):624-30.
- 42. Mucke M, Cuhls H, Radbruch L, Baron R, Maier C, Tolle T, et al. Quantitative sensory testing (QST). English version. Schmerz (Berlin, Germany). 2016.
- 43. De Groef A, Van Kampen M, Vervloesem N, Clabau E, Christiaens MR, Neven P, et al. Inter-rater reliability of shoulder measurements in middle-aged women. Physiotherapy. 2017;103(2):222-30.
- 44. Meeus M, Ickmans K, Struyf F, Hermans L, Van Noesel K, Oderkerk J, et al. Does acetaminophen activate endogenous pain inhibition in chronic fatigue syndrome/fibromyalgia and rheumatoid arthritis? A double-blind randomized controlled cross-over trial. Pain physician. 2013;16(2):E61-70.
- 45. Nahman-Averbuch H, Yarnitsky D, Granovsky Y, Sprecher E, Steiner M, Tzuk-Shina T, et al. Pronociceptive pain modulation in patients with painful chemotherapy-induced polyneuropathy. Journal of pain and symptom management. 2011;42(2):229-38.
- 46. Edwards RR, Mensing G, Cahalan C, Greenbaum S, Narang S, Belfer I, et al. Alteration in pain modulation in women with persistent pain after lumpectomy: influence of catastrophizing. Journal of pain and symptom management. 2013;46(1):30-42.

- 47. Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, et al. The Development and Psychometric Validation of the Central Sensitization Inventory. Pain Practice. 2012;12(4):276-85.
- 48. Scerbo T, Colasurdo J, Dunn S, Unger J, Nijs J, Cook C. Measurement Properties of the Central Sensitization Inventory: A Systematic Review. Pain Pract. 2017.
- 49. Cuesta-Vargas AI, Neblett R, Chiarotto A, Kregel J, Nijs J, van Wilgen CP, et al. Dimensionality and Reliability of the Central Sensitization Inventory in a Pooled Multicountry Sample. J Pain. 2018;19(3):317-29.
- 50. Lemmens RJ, Janssen-Potten YJ, Timmermans AA, Smeets RJ, Seelen HA. Recognizing complex upper extremity activities using body worn sensors. PloS one. 2015;10(3):e0118642.
- 51. Timmermans AA, Verbunt JA, van Woerden R, Moennekens M, Pernot DH, Seelen HA. Effect of mental practice on the improvement of function and daily activity performance of the upper extremity in patients with subacute stroke: a randomized clinical trial. Journal of the American Medical Directors Association. 2013;14(3):204-12.
- 52. Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011;63 Suppl 11:S174-88.
- 53. Sullivan M, Bishop S, Pivik J. The Pain Catastrophizing Scale: Development and Validation. Psychological Assessment. 1995;7(4):524-32.
- 54. Lovibond S, Lovibond P. Manual for the Depression Anxiety Stress Scales. Sydney: School of Psychology, University of New South Wales; 1995.
- 55. De Vrieze T, Coeck D, Verbelen H, Devoogdt N, Tjalma W, Gebruers N. Cross-cultural Psychometric Evaluation of the Dutch McGill-QoL Questionnaire for Breast Cancer Patients. Facts, views & vision in ObGyn. 2016;8(4):205-9.
- 56. Brouwer S, Franche R-L, Hogg-Johnson S, Lee H, Krause N, Shaw WS. Return-to-Work Self-Efficacy: Development and Validation of a Scale in Claimants with Musculoskeletal Disorders. Journal of occupational rehabilitation. 2011;21(2):244-58.
- 57. De Groef A, Van Kampen M, Vervloesem N, De Geyter S, Christiaens MR, Neven P, et al. Myofascial techniques have no additional beneficial effects to a standard physical therapy programme for upper limb pain after breast cancer surgery: a randomized controlled trial. Clinical rehabilitation. 2017:269215517708605.
- 58. De Groef A, Van Kampen M, Vervloesem N, Dieltjens E, Christiaens MR, Neven P, et al. Effect of myofascial techniques for treatment of persistent arm pain after breast cancer treatment: randomized controlled trial. Clinical rehabilitation. 2017:269215517730863.